CLINICAL TRIAL: NCT04247607
Title: A Prospective Observational Study of Patients Suffering From Prolonged Critical Illness Treated by Patient Centered Multidisciplinary Teams at a Specialized Unit: Patient Characteristics, Treatment and Follow-up Results
Brief Title: Specialized Treatment, Rehabilitation and Outcome in Patients With Prolonged Critical Illness
Acronym: CritillPro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Remeo AB (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2019120000; Dnr 2019-05294 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2020-01-02; First posted 2020-01-30 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Critical Illness
Keywords: persistent critical illness; chronic critical illness; prolonged intensive care; weaning from mechanical ventilation; decannulation; multidisciplinary team; intensive care rehabilitation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to describe the outcome for patients with persistent or chronic critical illness treated at Remeo, a clinic specialized for patients in need of prolonged intensive care and intensive care rehabilitation in Sweden. Patients' disease characteristics and the treatment in multidisciplinary patient centered teams for intensive care, weaning from mechanical ventilation and simultaneous rehabilitation will be described. Patients will be followed one year after discharge to document health related quality of life, physical function, frailty, mental illness and used health care resources.

ELIGIBILITY:
Inclusion Criteria:

Admission to unit (Remeo, Stockholm, Sweden) Treated for prolonged critical illness

Exclusion Criteria:

Treated less than 48 hours at unit (Remeo, Stockholm, Sweden)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with prolonged critical illness treated at the specialized unit (Remeo, Stockholm, Sweden)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in mechanical ventilation status | Assessed at admittance and immediately after discharge from unit
  Time (Days) from admittance to unit until weaned from mechanical ventilation
Change in tracheostomy status | Assessed at admittance and immediately after discharge from unit
  Time (Days) from admittance to unit until decannulation
In-patient mortality and mortality | Assessed immediately after discharge from unit
  Mortality during care at unit
Mortality during 12 months follow-up after discharge | Assessed 12 months after discharge
  Mortality during 12 months follow-up after discharge
Health related quality of Life assessed by the Rand 36-Item Health Survey (RAND36) | 3 months after discharge from unit
  RAND36 (scale 0-100, higher value better) questionnaire
Health related quality of Life assessed by the Rand 36-Item Health Survey (RAND36) | 6 months after discharge from unit
  RAND36 (scale 0-100, higher value better) questionnaire
Health related quality of Life assessed by the Rand 36-Item Health Survey (RAND36) | 12 months after discharge from unit
  RAND36 (scale 0-100, higher value better) questionnaire
Health related quality of Life assessed by EuroQoL 5-dimension 5-level (EQ-5D-5L) | 3 months after discharge from unit
  EQ-5D-5L questionnaire
Health related quality of Life assessed by EuroQoL 5-dimension 5-level (EQ-5D-5L) | 6 months after discharge from unit
  EQ-5D-5L questionnaire
Health related quality of Life assessed by EuroQoL 5-dimension 5-level (EQ-5D-5L) | 12 months after discharge from unit
  EQ-5D-5L questionnaire
Independence in activities of daily living assessed by Katz Index of Independence in Activities of Daily Living (Katz ADL) | At admission to unit
  Katz ADL (scale 0-6, higher value better)
Independence in activities of daily living assessed by Katz Index of Independence in Activities of Daily Living (Katz ADL) | Immediately before decannulation
  Katz ADL (scale 0-6, higher value better)
Independence in activities of daily living assessed by Katz Index of Independence in Activities of Daily Living (Katz ADL) | Immediately before discharge from unit
  Katz ADL (scale 0-6, higher value better)
Independence in activities of daily living assessed by Katz Index of Independence in Activities of Daily Living (Katz ADL) | 6 months after discharge from unit
  Katz ADL (scale 0-6, higher value better)
Independence in activities of daily living assessed by Katz Index of Independence in Activities of Daily Living (Katz ADL) | 12 months after discharge from unit
  Katz ADL (scale 0-6, higher value better)

SECONDARY OUTCOMES:
Symptoms of depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 3 months after discharge from unit
  PHQ-9, a patient related outcome questionnaire, scale 0-27, higher value indicating more severe symptoms
Symptoms of depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 6 months after discharge from unit
  PHQ-9, a patient related outcome questionnaire, scale 0-27, higher value indicating more severe symptoms
Symptoms of depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 12 months after discharge from unit
  PHQ-9, a patient related outcome questionnaire, scale 0-27, higher value indicating more severe symptoms
Symptoms of generalized anxiety as assessed by the General anxiety disorder 7 (GAD-7) questionnaire | 3 months after discharge from unit
  GAD-7, a patient related outcome questionnaire, scale 0-21, higher value indicating more severe symptoms
Symptoms of generalized anxiety as assessed by the General anxiety disorder 7 (GAD-7) questionnaire | 6 months after discharge
  GAD-7, a patient related outcome questionnaire, scale 0-21, higher value indicating more severe symptoms
Symptoms of generalized anxiety as assessed by the General anxiety disorder 7 (GAD-7) questionnaire | 12 months after discharge from unit
  GAD-7, a patient related outcome questionnaire, scale 0-21, higher value indicating more severe symptoms
Frailty as assessed by the Clinical frailty scale (CFS) | At admission to unit
  The Clinical frailty scale has 9 levels from very fit to terminally ill (1-9, lower value indicate better outcome)
Frailty as assessed by the Clinical frailty scale (CFS) | Immediately before discharge from unit
  The Clinical frailty scale has 9 levels from very fit to terminally ill (1-9, lower value indicate better outcome)
Frailty as assessed by the Clinical frailty scale (CFS) | At 6 months after discharge from unit
  The Clinical frailty scale has 9 levels from very fit to terminally ill (1-9, lower value indicate better outcome)
Frailty as assessed by the Clinical frailty scale (CFS) | At 12 months after discharge from unit
  The Clinical frailty scale has 9 levels from very fit to terminally ill (1-9, lower value indicate better outcome)
Physical status as assessed by the 6 minutes walk test | At admission to unit
  The 6 min walk test evaluated by a physiotherapist (longer distance (meters) better outcome)
Physical status as assessed by the 6 minutes walk test | Immediately before decannulation
  The 6 min walk test evaluated by a physiotherapist (longer distance (meters) better outcome)
Physical status as assessed by the 6 minutes walk test | Immediately before discharge from unit
  The 6 min walk test evaluated by a physiotherapist (longer distance (meters) better outcome)
Physical status as assessed by the 6 minutes walk test | 6 months after discharge from unit
  The 6 min walk test evaluated by a physiotherapist (longer distance (meters) better outcome)
Physical status as assessed by the 6 minutes walk test | 12 months after discharge from unit
  The 6 min walk test evaluated by a physiotherapist (longer distance (meters) better outcome)
Cognitive status as assessed by the Montreal cognitive assessment (MoCa) test | At admission to unit
  Performed by an occupational therapist. The MoCa test score scale is 0-30 Points, higher value indicate better outcome
Cognitive status as assessed by the Montreal cognitive assessment (MoCa) test | Immediately before decannulation
  Performed by an occupational therapist. The MoCa test score scale is 0-30 Points, higher value indicate better outcome
Cognitive status as assessed by the Montreal cognitive assessment (MoCa) test | Immediately before discharge from unit
  Performed by an occupational therapist. The MoCa test score scale is 0-30 Points, higher value indicate better outcome
Physical status as assessed by the Chelsea Critical Care Physical Assessment tool (CPAx). | At admission to unit
  CPAx performed by a physiotherapist (scale 0-50 Points, higher value indicate better outcome)
Physical status as assessed by the Chelsea Critical Care Physical Assessment tool (CPAx). | Immediately after decannulation
  CPAx performed by a physiotherapist (scale 0-50 Points, higher value indicate better outcome)
Physical status as assessed by the Chelsea Critical Care Physical Assessment tool (CPAx). | Immediately before discharge from unit
  CPAx performed by a physiotherapist (scale 0-50 Points, higher value indicate better outcome)
Physical status as assessed by the Chelsea Critical Care Physical Assessment tool (CPAx). | 6 months after discharge from unit
  CPAx performed by a physiotherapist (scale 0-50 Points, higher value indicate better outcome)
Physical status as assessed by the Chelsea Critical Care Physical Assessment tool (CPAx). | 12 months after discharge from unit
  CPAx performed by a physiotherapist (scale 0-50 Points, higher value indicate better outcome)
Swallowing function and possibility of oral intake | At admission to unit
  Using the Functional oral intake scale (FOIS)
Swallowing function and possibility of oral intake | Immediately before decannulation
  Using the Functional oral intake scale (FOIS)
Swallowing function and possibility of oral intake | Immediately before discharge from unit
  Using the Functional oral intake scale (FOIS), seven different levels 1-7, higher level indicate better function
Swallowing function and possibility of oral intake | At at 6 months after discharge from unit
  Using the Functional oral intake scale (FOIS), seven different levels 1-7, higher level indicate better function
Swallowing function and possibility of oral intake | At at 12 months after discharge from unit
  Using the Functional oral intake scale (FOIS), seven different levels 1-7, higher level indicate better function
Inflammatory status relative to outcome | Through study completion, an average of 14 months
  HMGB1 and routine inflammation markers' effect on outcome measures

OTHER OUTCOMES:
Antibiotic use | From admittance until discharge
  Days with antibiotic treatment during stay at unit.
Antibiotic use 12 months after discharge | From discharge until12 month thereafter
  Number of infections treated with antibiotics after discharge
Discharge destination | Immediately after discharge from unit
  The location the patient was discharged to; home, rehabilitation unit, acute care hospital, nursing home, palliative care unit
Need of support after discharge for patients discharged home | Immediately after discharge from unit
  For patients discharged home, the type of homecare needed (if any)
Number and type of Health care Contacts after discharge | Assessed 12 months after discharge from unit
  Number of Contacts with primary care, emergency room and hospital admissions after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eva Sundman, MD, PhD, Principal Investigator — Remeo and Karolinska Institutet
Locations (1):
- Remeo, Sköndal, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No